CLINICAL TRIAL: NCT03974594
Title: Single-Dose, Randomized, Open-Label, Two-Way Crossover Study to Evaluate the Bioequivalence of Trifluridine and Tipiracil Tablets in Colorectal Cancer Patients Under Fasting or Postprandial Conditions
Brief Title: Bioequivalence Study of Trifluridine and Tipiracil Tablets in Colorectal Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTTQ-TAS-102-I-02
Record Dates: First submitted 2019-05-31; First posted 2019-06-05 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Trifluridine; tipiracil; trifluridine tipiracil drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trifluridine and Tipiracil Tablets (Experimental)
  Interventions: Drug: Trifluridine and Tipiracil Tablets
- TAS-102 (Active Comparator)
  Interventions: Drug: TAS-102

INTERVENTIONS:
Drug: Trifluridine and Tipiracil Tablets — Trifluridine and Tipiracil Tablets given 20mg orally once under fasting or postprandial conditions per cycle
  Arms: Trifluridine and Tipiracil Tablets
Drug: TAS-102 — TAS-102 given 20mg orally once under fasting or postprandial conditions per cycle
  Arms: TAS-102

SUMMARY:
Trifluridine and Tipiracil Tablets is a nucleoside anti-metabolic and anti-cancer compound developed by Taiho (Dapeng) Co., Ltd., Japan, for the treatment of advanced colorectal cancer that inoperable resection, and progressed or relapsed after standard treatment. This study mainly evaluates bioequivalence, safety and tolerance of Trifluridine and Tipiracil Tablets in colorectal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. 18-70 years old, life expectancy ≥ 3 months.
2. Histologically confirmed colon or rectal adenocarcinoma.
3. Has not received anti-tumor therapy before 4 weeks of first dose or Traditional Chinese Medicine anti-tumor therapy before 2 weeks of first dose.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
5. Has ability to take oral medication.
6. The main organs function are normally, the following criteria are met:

   1. Hemoglobin (HB) ≥ 100 g / L;
   2. Absolute neutrophil count (ANC) ≥1.5×109/L;
   3. Platelets (PLT) ≥ 80 × 109 / L;
   4. Total serum bilirubin (TBIL) ≤ 1.5 × ULN;
   5. Alanine transaminase (ALT) and Aspartate aminotransferase (AST) ≤ 2.5 × ULN (when the liver is invaded，AST ≤ 5×ULN);
   6. Serum creatinine ≤ 132.6 μmol / L.
7. Male or female subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 6 months after the last dose of study (such as intrauterine devices , contraceptives or condoms) ；No pregnant or breastfeeding women, and a negative pregnancy test are received within 7 days before the randomization.
8. Understood and signed an informed consent form.

Exclusion Criteria:

1. Has serious diseases , including but not limited to:

   1. Has diagnosed and/or treated additional malignancy within 5 years prior to randomization. Exceptions include carcinoma in situ of cervix, non-melanoma skin cancer and superficial bladder tumor;
   2. Has brain metastases;
   3. Has active infection (such as infection caused body temperature ≥ 38 ° C);
   4. Has pleural effusion, pericardial effusion, or ascites requiring recurrent drainage before 4 weeks of first dose;
   5. Has intestinal obstruction, pulmonary fibrosis, renal failure, liver failure or symptomatic cerebrovascular disease;
   6. Has uncontrolled diabetes (fasting blood glucose (FBG) > 10mmol/L);
   7. Has myocardial infarction, severe/unstable angina pectoris, New York Heart Association (NYHA) grade III or IV symptomatic congestive heart failure within 12 months prior to first dose;
   8. Has gastrointestinal bleeding;
   9. Has HIV infection, or active hepatitis B or C;
   10. Has a history of organ transplants or autoimmune disease required immunosuppressive therapy;
   11. Has increased risk associated with participating in the study or taking the study drug, or mental disorders may interfere with the results of the study.
2. Has received any of the following treatments before the first dose:

   1. Has received partial or total gastrectomy;
   2. Has surgery (such as laparotomy, thoracotomy, and laparoscopic resection of the viscera and/or unhealed wounds) within 4 weeks;
   3. Has any study drug within 4 weeks.
3. Prior therapy with TAS-102.
4. Has adverse events caused by previous therapy except alopecia that did not recover to ≤ grade 2.
5. Pregnant or lactating woman.
6. Subjects who, in the opinion of the investigators, should not participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2019-07-16 (Actual); Study Completion 2019-07-16 (Actual)

PRIMARY OUTCOMES:
AUC(0-infinity) | 3 days
  The AUC(0-infinity) is area under the serum concentration-time curve from time zero to infinite time.
AUC(0-t) | 3 days
  The AUC(0-t) is area under the serum concentration-time curve from time zero to t.
Bioequivalence based on Peak Plasma Concentration (Cmax) | 3 days
  The Cmax is observed maximum serum concentration, taken directly from the serum concentration-time profile

SECONDARY OUTCOMES:
Adverse Event | Up to 4 weeks
  Security Index

CONTACTS AND LOCATIONS:
Locations (1):
- Tangdu Hospital,Fourth Military Medical University, Xi’an, Shanxi, China

REFERENCES:
- [Derived] Su HC, Min J, Song Y, Liu LL, Liu LN, Zhang HL. A bioequivalence study of trifluridine/tipiracil tablets in Chinese metastatic colorectal cancer patients under fed conditions. Cancer Chemother Pharmacol. 2023 Feb;91(2):167-177. doi: 10.1007/s00280-022-04501-8. Epub 2023 Jan 9. PMID 36622402